#### TITLE PAGE

**Protocol Title:** A Randomized, Open-Label, Single Dose, Four-Period Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants

**Protocol Number**: 209713

Compound Number: GSK3640254

Study Phase: Phase 1

**Short Title:** A Relative Bioavailability and Food-Effect Study of GSK3640254 Tablet and Capsule Formulations in Healthy Participants

#### US IND Sponsor Name and Legal Registered Address:

ViiV Healthcare Company
Five Moore Drive
P.O. 13398
Research Triangle Park, NC 27709-3398, USA
Telephone: PPD

In some countries, local law requires that the Clinical Trial sponsor is a local company legal entity. In these instances, the appropriate company to be identified as Sponsor must be agreed with the global ViiV Healthcare clinical team and signed off by the Vice President, Global Research and Medical Strategy

This study is sponsored by ViiV Healthcare. PPD with GlaxoSmithKline are supporting ViiV Healthcare in the conduct of this study.

**Medical Monitor Name and Contact Information:** Can be found in the Study Reference Manual

**Regulatory Agency Identifying Number(s):** 

IND: 139,838

**Approval Date: 30-AUG-2019** 

Copyright 2019 the ViiV Healthcare group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

# **SPONSOR SIGNATORY:**

| r :ailiade, DO, MPH V1, cimical Development ViiV Healthcare | 8/30/20/9<br>Date |
|---|---|
| PPD | |

# **TABLE OF CONTENTS**

| 1. PROTOCOL SUMMARY 6 1.1. Synopsis 6 1.2. Schema 8 1.3. Schedule of Activities (SoA) 9 2. INTRODUCTION 13 2.1. Study Rationale 13 2.2. Background 13 2.2.1. Background and Key Safety Data With a Prior Maturation Inhibitor 13 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 15 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 16 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 20 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5.1 Inclusion Criteria 23 5.2 Exclusion Criteria 24 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity < | | | | PAGE |
|---|---|---|---|---|
| 1.1. Synopsis 6 1.2. Schema 8 1.3. Schedule of Activities (SoA) 9 2. INTRODUCTION 13 2.1. Study Rationale 13 2.2. Background and Key Safety Data With a Prior Maturation Inhibitor 13 1.1. Discontinuation 13 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 15 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 16 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria | 1. | PRO1 | FOCOL SUMMARY | 6 |
| 1.3. Schedule of Activities (SoA) | | | | |
| 2. INTRODUCTION | | 1.2. | | |
| 2.1. Study Rationale 13 2.2. Background 13 2.2.1. Background and Key Safety Data With a Prior Maturation Inhibitor 13 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 15 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 17 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.2. | | 1.3. | Schedule of Activities (SoA) | 9 |
| 2.1. Study Rationale 13 2.2. Background 13 2.2.1. Background and Key Safety Data With a Prior Maturation Inhibitor 13 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 15 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 17 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.2. | 2 | INTR | ODLICTION | 13 |
| 2.2.1 Background and Key Safety Data With a Prior Maturation Inhibitor. 13 2.2.1. Background and Key Safety Data With a Prior Maturation Inhibitor. 13 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187. 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131. 15 2.3. Benefit/Risk Assessment. 16 2.3.1. Risk Assessment. 17 2.3.2. Benefit Assessment. 20 2.3.3. Overall Benefit: Risk Conclusion. 20 3. OBJECTIVES AND ENDPOINTS. 20 4. STUDY DESIGN. 20 4.1. Overall Design. 20 4.2. Scientific Rationale for Study Design. 21 4.3. Justification for Dose. 22 4.4. End-of-Study Definition. 22 5. STUDY POPULATION. 22 5.1. Inclusion Criteria. 23 5.2. Exclusion Criteria. 24 5.3.1. Meals and Dietary Restrictions. 26 5.3.1. Meals and Dietary Restrictions. 26 5.3.2. <t< td=""><td>۷.</td><td></td><td></td><td></td></t<> | ۷. | | | |
| 2.2.1 Background and Key Safety Data With a Prior Maturation Inhibitor | | | | |
| 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187 14 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 15 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 17 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 20 20 20 20 20 20 2 | | ۷.۷. | 2.2.1. Background and Key Safety Data With a Prior Maturation | |
| 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131 | | | 2.2.2. Preliminary Safety and Pharmacokinetic Data in | |
| 2.3. Benefit/Risk Assessment 16 2.3.1. Risk Assessment 17 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Faillures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study | | | 2.2.3. Preliminary Safety and Pharmacokinetic Data in | |
| 2.3.1. Risk Assessment 20 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION A | | 23 | | |
| 2.3.2. Benefit Assessment 20 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION WITHDRAWAL 29 | | 2.0. | | |
| 2.3.3. Overall Benefit: Risk Conclusion 20 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 </td <td></td> <td></td> <td></td> <td></td> | | | | |
| 3. OBJECTIVES AND ENDPOINTS 20 4. STUDY DESIGN 20 4.1. Overall Design 21 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | | | |
| 4. STUDY DESIGN 20 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | | | 20 |
| 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | 3. | OBJE | CTIVES AND ENDPOINTS | 20 |
| 4.1. Overall Design 20 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | 4. | STUD | DY DESIGN | 20 |
| 4.2. Scientific Rationale for Study Design 21 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6. STUDY INTERVENTION 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | | | |
| 4.3. Justification for Dose 22 4.4. End-of-Study Definition 22 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | 4.2. | <u> </u> | |
| 5. STUDY POPULATION 22 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | 4.3. | | |
| 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | | 4.4. | End-of-Study Definition | 22 |
| 5.1. Inclusion Criteria 23 5.2. Exclusion Criteria 24 5.3. Lifestyle Considerations 26 5.3.1. Meals and Dietary Restrictions 26 5.3.2. Caffeine, Alcohol, and Tobacco 27 5.3.3. Activity 27 5.4. Screen Failures 27 6.1. Study Interventions Administered 28 6.2. Preparation/Handling/Storage/Accountability 28 6.3. Measures to Minimize Bias: Randomization and Blinding 29 6.4. Study Intervention Compliance 29 6.5. Concomitant Therapy 29 6.6. Dose Modification 29 6.7. Intervention After the End of the Study 29 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL 29 7.1. Discontinuation of Study Intervention 29 | 5. | STUD | OY POPULATION | 22 |
| 5.2. Exclusion Criteria245.3. Lifestyle Considerations265.3.1. Meals and Dietary Restrictions265.3.2. Caffeine, Alcohol, and Tobacco275.3.3. Activity275.4. Screen Failures276. STUDY INTERVENTION276.1. Study Interventions Administered286.2. Preparation/Handling/Storage/Accountability286.3. Measures to Minimize Bias: Randomization and Blinding296.4. Study Intervention Compliance296.5. Concomitant Therapy296.6. Dose Modification296.7. Intervention After the End of the Study297. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL297.1. Discontinuation of Study Intervention29 | | | | |
| 5.3.1. Meals and Dietary Restrictions | | _ | | |
| 5.3.1. Meals and Dietary Restrictions | | 5.3. | Lifestyle Considerations | 26 |
| 5.3.3. Activity | | | | |
| 5.4. Screen Failures | | | 5.3.2. Caffeine, Alcohol, and Tobacco | 27 |
| 5.4. Screen Failures | | | 5.3.3. Activity | 27 |
| 6.1. Study Interventions Administered286.2. Preparation/Handling/Storage/Accountability286.3. Measures to Minimize Bias: Randomization and Blinding296.4. Study Intervention Compliance296.5. Concomitant Therapy296.6. Dose Modification296.7. Intervention After the End of the Study297. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL297.1. Discontinuation of Study Intervention29 | | 5.4. | | |
| 6.1. Study Interventions Administered286.2. Preparation/Handling/Storage/Accountability286.3. Measures to Minimize Bias: Randomization and Blinding296.4. Study Intervention Compliance296.5. Concomitant Therapy296.6. Dose Modification296.7. Intervention After the End of the Study297. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL297.1. Discontinuation of Study Intervention29 | 6 | STUE | OY INTERVENTION | 27 |
| 6.2.Preparation/Handling/Storage/Accountability286.3.Measures to Minimize Bias: Randomization and Blinding296.4.Study Intervention Compliance296.5.Concomitant Therapy296.6.Dose Modification296.7.Intervention After the End of the Study297.DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL297.1.Discontinuation of Study Intervention29 | ٥. | | | |
| 6.3. Measures to Minimize Bias: Randomization and Blinding | | | | |
| 6.4. Study Intervention Compliance | | | | |
| 6.5. Concomitant Therapy | | | | |
| 6.6. Dose Modification | | | | |
| 6.7. Intervention After the End of the Study | | | | |
| DISCONTINUATION/WITHDRAWAL | | | | |
| DISCONTINUATION/WITHDRAWAL | 7 | DISC | ONTINUATION OF STUDY INTERVENTION AND PARTICIPANT | |
| 7.1. Discontinuation of Study Intervention | ٠. | | | 20 |

| | | 7.1.1.1. Study Intervention Restart or Rechallenge After | 00 |
|---|---|---|---|
| | | Liver Stopping Criteria Met | |
| | | 7.1.2. QTc Stopping Criteria | 30 |
| | | 7.1.3. Columbia Suicide Severity Rating Scale Criteria | 30 |
| | | 7.1.4. Individual Participant Laboratory Abnormality and Adverse | 24 |
| | 7.2. | Event Stopping Criteria | 31 |
| | 7.2.<br>7.3. | Participant Discontinuation/Withdrawal From the StudyLost to Follow-Up | |
| | 1.3. | Lost to Follow-op | 32 |
| 8. | STUD | Y ASSESSMENTS AND PROCEDURES | 32 |
| | 8.1. | Efficacy Assessments | |
| | 8.2. | Safety Assessments | |
| | | 8.2.1. Physical Examinations | 33 |
| | | 8.2.2. Vital Signs | 33 |
| | | 8.2.3. Electrocardiograms | 33 |
| | | 8.2.4. Clinical Safety Laboratory Assessments | 34 |
| | | 8.2.5. Suicidal Risk Monitoring and Management of Emergent | |
| | | Psychiatric Symptoms | |
| | | 8.2.6. Gastrointestinal Toxicity Evaluation and Monitoring Plan | |
| | 8.3. | Adverse Events and Serious Adverse Events | 37 |
| | | 8.3.1. Time Period and Frequency for Collecting AE and SAE | |
| | | Information | 37 |
| | | 8.3.2. Method of Detecting AEs and SAEs | |
| | | 8.3.3. Follow-up of AEs and SAEs | |
| | | 8.3.4. Regulatory Reporting Requirements for SAEs | |
| | 0.4 | 8.3.5. Pregnancy | |
| | 8.4. | Treatment of Overdose | |
| | 8.5. | Pharmacokinetics | |
| | 8.6.<br>8.7. | Pharmacodynamics | |
| | 6.7.<br>8.8. | Genetics Biomarkers | |
| | 8.9. | Medical Resource Utilization and Health Economics | |
| | 0.9. | Wedical Resource Offitzation and Health Economics | 40 |
| 9. | STAT | ISTICAL CONSIDERATIONS | 40 |
| | 9.1. | Statistical Hypotheses | 40 |
| | 9.2. | Sample Size Determination | 40 |
| | | 9.2.1. Sample Size Assumptions | 40 |
| | | 9.2.2. Sample Size Sensitivity | |
| | 9.3. | Populations for Analyses | |
| | 9.4. | Statistical Analyses | |
| | | 9.4.1. Pharmacokinetic Analyses | |
| | | 9.4.2. Safety Analyses | |
| | | 9.4.3. Other Analyses | |
| | 9.5. | Interim Analyses | |
| | | 9.5.1. Data Monitoring Committee (DMC) | 44 |
| 10 | SLIDD | ORTING DOCUMENTATION AND OPERATIONAL | |
| ıυ. | | SIDERATIONS | 15 |
| | 10.1. | | |
| | 10.1. | Appendix 2: Clinical Laboratory Tests | |
| | 10.2. | • • | |
| | | Information | 50 |

| | | 10.3.1. Definitions | 50 |
|----|-------|------------------------------------------------------------|----|
| | | 10.3.1. Collection of Pregnancy Information | |
| | 10.4. | Appendix 4: Regulatory, Ethical, and Study Oversight | |
| | | Considerations | 53 |
| | | 10.4.1. Regulatory and Ethical Considerations | 53 |
| | | 10.4.2. Financial Disclosure | |
| | | 10.4.3. Informed Consent Process | |
| | | 10.4.4. Data Protection | |
| | | 10.4.5. Publication Policy | |
| | | 10.4.6. Dissemination of Clinical Study Data | |
| | | 10.4.7. Data Quality Assurance | |
| | | 10.4.8. Source Documents | |
| | | 10.4.9. Study and Site Closure | 56 |
| | 10.5. | Appendix 5: Liver Safety: Required Actions and Follow-up | |
| | | Assessments | 57 |
| | 10.6. | Appendix 6: Adverse Events: Definitions and Procedures for | |
| | | Recording, Evaluating, Follow-up, and Reporting | 59 |
| | | 10.6.1. Definition of AE | |
| | | 10.6.2. Definition of SAE | |
| | | 10.6.3. Recording and Follow-Up of AE and SAE | 61 |
| | | 10.6.4. Reporting of SAE to VH/GSK | |
| | 10.7. | · | |
| 11 | RFFF | RENCES | 65 |

#### 1. PROTOCOL SUMMARY

# 1.1. Synopsis

**Protocol Title:** A Randomized, Open-Label, Single Dose, Four-Period Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants

**Short Title:** A Relative Bioavailability and Food-Effect Study of GSK3640254 Tablet and Capsule Formulations in Healthy Participants

#### Rationale:

This is an open-label, single-dose, 4-period crossover study to compare the relative bioavailability (BA) of the GSK3640254 formulation planned for Phase 2b (mesylate salt in a tablet) with the Phase 2a formulation (mesylate salt in a capsule) when administered following a moderate calorie and fat meal. Data from this study will determine whether dose adjustments are required due to formulation changes when transitioning from Phase 2a to Phase 2b clinical studies.

In addition, this study will investigate the effect of food on the pharmacokinetics (PK) of the GSK3640254 mesylate tablet formulation. All GSK3640254 clinical studies to date, including a Phase 2a proof of concept study, have been conducted with moderate calorie and fat meals. It is intended that this will be the only food-effect BA clinical study for GSK3640254; therefore, this study will investigate the effect of moderate and high calorie and fat meals on the PK, safety, and tolerability of the GSK3640254 mesylate tablet formulation, as compared to administration under fasting conditions.

#### **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the relative bioavailability of<br>GSK3640254 mesylate tablets and<br>GSK3640254 mesylate capsules (in the<br>presence of a moderate fat meal) | AUC(0-∞), AUC(0-t), Cmax, and Tmax for<br>GSK3640254 |
| To assess the effect of food (fasted,<br>moderate fat meal, and high fat meal) on<br>the PK of the GSK3640254 mesylate tablet<br>formulation | |

| Objectives | Endpoints |
|---|---|
| Secondary | |
| To assess the safety and tolerability of<br>GSK3640254 following single oral<br>administration to healthy participants under<br>fasted or fed (moderate fat or high fat)<br>conditions | Safety and tolerability parameters for<br>AEs/SAEs, observed and change from<br>Baseline clinical laboratory assessments,<br>ECGs, and vital sign measurements |
| To characterize the PK of GSK3640254 | <ul> <li>tlag, t1/2, CL/F, and Vz/F for GSK3640254</li> <li>GSK3640254 PK concentrations in plasma</li> </ul> |

AE = adverse event;  $AUC(0-\infty)$  = area under the plasma concentration-time curve from time zero extrapolated to infinity; AUC(0-t) = area under the plasma concentration-time curve from time zero to time t; CL/F = apparent oral clearance; Cmax = maximum observed concentration; ECG = electrocardiogram; PK = pharmacokinetics; SAE = serious adverse event; t1/2 = apparent terminal phase half-life; tlag = lag time for absorption; Tmax = time of maximum observed concentration; Vz/F = apparent volume of distribution.

#### **Overall Design:**

This is a Phase 1, randomized, open-label, single-dose, 4-period crossover study to compare the relative BA of a tablet formulation of GSK3640254 with the capsule formulation and to assess the effect of food on the PK of the tablet formulation in healthy participants.

The study will consist of a Screening period and 4 sequential treatment periods with a single dose of study intervention per treatment period.

For treatments administered in the fed state, participants will fast overnight for at least 10 hours prior to dosing and will receive a moderate fat or high fat meal 30 minutes prior to dosing. Dose administration will occur within 5 minutes of completion of meal consumption. Participants will not receive any further food until 4 hours after dosing. For treatments administered in the fasted state, participants will fast overnight for at least 10 hours prior to dosing and until 4 hours after dosing.

Pharmacokinetic blood samples for the analysis of GSK3640254 will be collected prior to dosing (0 hour) on Day 1 and up to 96 hours postdose in Periods 1, 2, 3, and 4.

Safety and tolerability will be assessed by monitoring and recording of adverse events, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram results, and physical examination findings.

Study assessments will be performed as indicated in the Schedule of Activities (Section 1.3). Study participants will be confined to the clinic from Day –1 until discharge on Day 5 of Period 4.

**Disclosure Statement**: This is a crossover treatment study with 1 arm that has no masking.

**Number of Participants:** Approximately 16 participants will be treated to ensure that 12 evaluable participants complete the study. If participants prematurely discontinue the study, additional participants may be randomized after consultation with the sponsor to ensure that 12 evaluable participants complete the study.

**Intervention Groups and Duration:** Prior to dosing on Day 1 of Period 1, participants will be randomly assigned to 1 of 4 treatment sequences (ABCD, BADC, CDAB, or DCBA). Participants will receive each of the following treatments administered as 1 treatment per period:

- Treatment A: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg capsules) administered under moderate fat conditions (reference).
- Treatment B: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under moderate fat conditions (test).
- Treatment C: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under fasted conditions (reference).
- Treatment D: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under high fat conditions (test).

To ensure adequate washout, there will be at least 7 days between each dose of study intervention, with an allowance window of 4 hours (i.e., 7 days minus 4 hours) to allow flexibility in scheduling participants for dosing at the clinic. The duration of the study, including Screening, is approximately 54 days.

**Data Monitoring Committee: No** 

#### 1.2. Schema

A summary of the overall study design is presented in Figure 1.

Figure 1 Study Design Schematic



Treatment A = GSK3640254 200 mg (capsules) administered under moderate fat conditions;

Treatment B = GSK3640254 200 mg (tablets) administered under moderate fat conditions;

Treatment C = GSK3640254 200 mg (tablets) administered under fasted conditions;

Treatment D = GSK3640254 200 mg (tablets) administered under high fat conditions.

1 Washout will be at least 7 days minus 4 hours.

# 1.3. Schedule of Activities (SoA)

- Screening procedures may be done over more than 1 visit but must all be completed within 28 days prior to the first dose of study intervention.
- The following demographic parameters will be captured: year of birth, sex, race, and ethnicity.
- Medical/medication/family history will be assessed as related to the inclusion/exclusion criteria.

# **Screening Visit**

| Procedure | Screening (up to 28 days before Day 1) |
|---|---|
| Outpatient visit | X |
| Informed consent | X |
| Inclusion and exclusion criteria | X |
| Demography | X |
| Full physical examination including height and weight 1 | Х |
| Laboratory assessments (hematology, chemistry, urinalysis) | X |
| 12-lead electrocardiogram | X |
| Vital sign measurements | Х |
| Medication/drug/alcohol history | X |
| Past and current medical conditions | X |
| Columbia Suicide Severity Rating Scale | X |
| Serum pregnancy test | X |
| Follicle-stimulating hormone (as needed, to confirm postmenopausal status) | X |
| Drug, alcohol, and cotinine screen | Х |
| Human immunodeficiency virus, hepatitis B and C Screening | Х |

<sup>1</sup> A full physical examination will include at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal, and neurological systems.

## **Time and Events Table**

| Procedure | Check-in | | Periods | 1, 2, and 3 | 3 | Period 4 only | | | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|
| | _ | _ | | Washout | | _ | _ | _ | _ | |
| | Day<br>-1 | Day<br>1 | Day<br>2 | Days<br>3-5 | Days<br>6-7 | Day<br>1 | Day<br>2 | Days<br>3-4 | Day<br>5 <sup>1</sup> | |
| Admit to clinic | Х | | | | | | | | | |
| Discharge from clinic | | | | | | | | | Х | Discharge from clinic following completion of the last study procedure on Day 5 of Period 4. |
| Brief physical examination | Х | | | | D7<br>(Period 2<br>only) | | | | X | Interim or symptom targeted physical examination will be performed at the discretion of the investigator. See Section 8.2.1 for description of brief physical examination. |
| Vital signs | х | Х | Х | D3-5 | | Х | Х | х | Х | Blood pressure and pulse will be measured in triplicate predose on Day 1 in Periods 1-4. Single blood pressure and pulse will be measured predose on other study days. |
| 12-lead ECG | х | Х | | | | Х | | | Х | All ECGs on Day 1 in Periods 1-4 will be predose, postdose at 2 hours, and postdose at 4 hours. The predose ECGs in Periods 1-4 will be taken in triplicate. |
| Drug, alcohol, and cotinine screen | Х | | | | | | | | | See Appendix 2 for specific tests to be performed. |
| Laboratory<br>assessments<br>(hematology, chemistry,<br>urinalysis) | Х | | Х | | | | Х | | Х | See Appendix 2 for specific tests to be performed. Day 2 samples in each period to be collected 24 hours after dosing. |

| Procedure | Check-in | | Periods 1, 2, and 3 | | | Period 4 only | | | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Davi | Davi | | Washou | t | Davi | Dovi | Davis | _ | |
| | Day<br>-1 | Day<br>1 | Day<br>2 | Days<br>3-5 | Days<br>6-7 | Day<br>1 | Day<br>2 | Days<br>3-4 | Day<br>5 <sup>1</sup> | |
| Pregnancy test | Х | | | | | | | | Χ | Serum testing at Day -1 |
| Columbia-Suicide<br>Severity<br>Rating Scale | Х | | | | D7 | | | | Х | |
| Genetic sample (optional) | Х | | | | | | | | | |
| Study intervention:<br>GSK3640254 200 mg<br>(capsule or tablet) | | Х | | | | х | | | | Participants will fast overnight for at least 10 hours prior to dosing; be provided a moderate fat meal, a high fat meal, or no meal 30 minutes prior to dosing; and be provided standardized meals ≥4 hours postdose. See Section 4.1. |
| Serial PK sampling | | Х | Х | Х | | Х | Х | х | Х | Blood collection for PK analysis of GSK3640254 will be collected within 40 minutes prior to dosing and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose in each period. |
| AE review | | ← | | | | | | <b>&gt;</b> | | |
| SAE review | <b>←===</b> | ← | | | | | | <del>}</del> | | |
| Concomitant medications | <b>←</b> =======X======X=======→ | | | | | | | | | |

AE = adverse event; D = day; ECG = electrocardiogram; PK = pharmacokinetic; SAE = serious adverse event.

1 Evaluations scheduled for Day 5 in Period 4 will also be performed for participants who discontinue early.

2018N383392\_00 **CONFIDENTIAL** 209713

• The timing and number of planned study assessments, including safety, PK, or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

• Any changes in the timing or addition of time points for any planned study assessments as the result of emerging PK data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files but will not constitute a protocol amendment. The Institutional Review Board/Independent Ethics Committee will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the informed consent form. The changes will be approved by the competent authorities and the ethics committee before implementation.

#### 2. INTRODUCTION

# 2.1. Study Rationale

This is an open-label, single-dose, 4-period crossover study to compare the relative bioavailability (BA) of the GSK3640254 formulation planned for Phase 2b (mesylate salt in a tablet) with the Phase 2a formulation (mesylate salt in a capsule) when administered following a moderate calorie and fat meal. Data from this study will determine whether dose adjustments are required due to formulation changes when transitioning from Phase 2a to Phase 2b clinical studies.

In addition, this study will investigate the effect of food on the pharmacokinetics (PK) of the GSK3640254 mesylate tablet formulation. All GSK3640254 clinical studies to date, including a Phase 2a proof of concept study, have been conducted with moderate calorie and fat meals. It is intended that this will be the only food-effect BA clinical study for GSK3640254; therefore, this study will investigate the effect of moderate and high calorie and fat meals on the PK, safety, and tolerability of the GSK3640254 mesylate tablet formulation, as compared to administration under fasting conditions.

## 2.2. Background

GSK3640254 is a human immunodeficiency virus (HIV) maturation inhibitor (MI) which is improved over prior developmental MIs in the following ways: (1) it exhibits significantly improved pan-genotypic coverage and potency against polymorphic variants; (2) *in vitro* data suggest that GSK3640254 exhibits a higher barrier to emergence of resistant viruses (except for A364V); (3) GSK3640254 has improved potency *in vitro* toward all HIV-1 subtypes; (4) it has potential for improved gastrointestinal (GI) tolerability; and (5) it has a projected lower once-daily human dose. Summaries of the pre-clinical and clinical studies are included in the Clinical Investigator's Brochure (CIB) [GlaxoSmithKline (GSK) Document Number 2018N379610 00].

# 2.2.1. Background and Key Safety Data With a Prior Maturation Inhibitor

Bristol-Myers Squibb (BMS), and later ViiV Healthcare (VH), developed a structurally similar HIV-1 MI (BMS-955176/GSK3532795), which was studied through Phase 2b studies in both treatment-naïve (AI468038/205891) and experienced (AI468048/205892) HIV-1 infected adults. In study AI468038/205891, a greater number of participants who received GSK3532795 experienced GI intolerability (most frequently Grade 1 to 2 diarrhea and abdominal pain). A detailed examination of all GI adverse events (AEs) (regardless of grade/relationship) revealed a relationship with dose [GSK Document Number 2016N302783\_00]. Ultimately, the rate of GI intolerability in the GSK3532795 dose groups in the Phase 2b study 205891 led to VH's decision to end all trials and not progress to Phase 3 studies. Gastrointestinal AEs were also previously observed in healthy participants in Phase 1 studies with varying doses, durations, and formulations of GSK3532795. In all 3 studies, the most common GI AEs were abdominal pain and diarrhea.

Aside from mild to moderate GI intolerability, 2 serious adverse events (SAEs) occurred in the Phase I thorough QT study AI468044/206220 [BMS Document Control Number 930109388] at supra-therapeutic doses: 1 healthy participant had an episode of acute psychosis and another had suicidal ideation/homicidal ideation as diagnosed through an interview by a psychiatrist. The 2 participants received GSK3532795 240 mg twice daily and 240 mg once daily (QD) with food, respectively. These events were assessed as related to study intervention but were not observed in any other clinical study with GSK3532795. The most frequent neuropsychiatric AEs in studies with GSK3532795 were headache, dizziness, and sleep abnormalities (e.g., insomnia, abnormal dreams).

# 2.2.2. Preliminary Safety and Pharmacokinetic Data in Study 207187

The primary objective of the first time in human (FTIH) clinical trial (207187) was to investigate the safety and tolerability of GSK3640254 following single and repeated daily administration. A total of 78 healthy men were ultimately randomized: 20 in the single-ascending dose ([SAD], doses ranging from 1 to 700 mg) and 58 in the multiple-ascending dose ([MAD], 50 to 320 mg QD for 14 days). A comprehensive summary of results is described in the CIB [GSK Document Number 2018N379610\_00] and the Study Synopsis [GSK Document Number 2018N375461\_00]. A concise summary of the data is presented below.

No deaths or SAEs were reported. There were 4 AEs leading to discontinuation. Only 1 of these AEs was related to study medication. A participant who received GSK3640254 200 mg QD developed a maculopapular rash after 8 days of study medication. The rash lasted for 6 days and there were no laboratory abnormalities. A dermatology consultant concluded this was a drug rash and the participant later received fexofenadine 180 mg QD and a topical steroid cream with resolution of the rash. The other 3 AEs occurred in SAD portion of the study (depression in a participant who received placebo and 2 participants with viral infection).

There were 9 participants with 12 AEs assessed as related to study medication by the principal investigator (11 Grade 1; 1 Grade 2). The most clinically notable was a participant who developed elevated transaminases while receiving GSK3640254 50 mg QD for 14 days. Specifically, there was a progressive rise in alanine aminotransferase (ALT) during treatment with a peak ALT of 83 IU/L on Day 16. The remaining liver chemistries were normal throughout. An ultrasound showed a subcapsular area of heterogenous echogenicity within segment 7, measuring approximately 35 × 23 × 36 mm. Follow-up magnetic resonance imaging and liver chemistries were normal. This participant also had 3 unrelated AEs during the course of an isolated increased ALT: musculoskeletal stiffness, contact dermatitis, and headache. All other related AEs are described in the CIB) [GSK Document Number 2018N379610\_00] and the Study Synopsis [GSK Document Number 2018N375461\_00].

In the SAD portion of the study, 17 participants experienced 60 individual AEs (58 Grade 1; 2 Grade 2). The 2 Grade 2 AEs were headache and depression (both unrelated). The most frequent AEs were headache, contact dermatitis primarily due to electrocardiogram (ECG) electrodes, and diarrhea. There was no dose/AE relationship.

In the MAD portion of the study, 44 participants experienced 130 individual AEs (126 Grade 1; 4 Grade 2). The 4 Grade 2 AEs were headache (1 related and 1 unrelated) and back pain (2 unrelated). The most frequent AEs were headache, contact dermatitis, dizziness, contusion, fatigue, and back pain.

There were no clinically significant abnormal fluctuations or trends in vital signs in the SAD or MAD cohorts. There were no abnormal clinically significant arrhythmias or QT prolongations (values >500 ms or increases >60 ms from Baseline) observed for any participant in the SAD or MAD. A cardiodynamic evaluation of healthy participants in the MAD portion of Study 207187 (placebo or GSK3640254 dose range 50 to 320 mg daily for 14 days) was performed. Serial ECGs were extracted from continuous Holter monitors at time-matched Baseline on Day -1 and for approximately 24 hours post-dose on Days 1 and 14. In the concentration-corrected OT interval (OTc) analysis, a final model with a treatment effect-specific intercept reasonably represented the data. The slope of the concentration-QTc relationship was 0.004 ms per ng/mL (90% confidence interval [CI]: 0.0023 to 0.0048) with a small treatment effect-specific intercept of -0.9 ms (90% CI: -4.47 to 2.69). The QT effect ( $\Delta\Delta$ QTcF) of GSK3640254 could be predicted to be 5.38 ms (90% CI: 1.66 to 9.10) and 6.70 ms (90% CI: 2.79 to 10.61) for the 200 mg (1779 ng/mL) and 320 mg (2154 ng/mL) doses, respectively, on Day 14. Based on this concentration-QTc analysis, a QTc using the Fridericia formula (QTcF) effect above 10 ms could be excluded up to GSK3640254 plasma concentrations of approximately 2000 ng/mL (corresponding to doses approximately ≤200 mg QD; note, the dose used in this study is 200 mg QD). Finally, there were no laboratory abnormality trends across doses that were clinically significant or associated with any symptoms.

Preliminary GSK3640254 PK parameters derived based on nominal sampling times following single doses of 1 to 700 mg administered after a moderate calorie and fat breakfast showed GSK3640254 was slowly absorbed with a median time of maximum observed concentration (Tmax) observed between 3 to 4.5 hours after dosing with a moderate fat breakfast and slowly eliminated with a mean half-life ranging from 22 to 26 hours. In general, exposure (maximum observed concentration [Cmax] and area under the plasma concentration-time curve [AUC]) increased in a close-to-dose-proportional manner from 1 to 400 mg with no further increase in exposure at 700 mg.

Repeat dose preliminary PK parameters following administration of GSK3640254 50 to 320 mg QD for 14 days were determined on Day 1 and Day 14 and showed a median Tmax ranging from 3.8 to 4.3 hours. The mean half-life ranged from approximately 22 to 29 hours. Overall, there was a trend of a slightly less than dose-proportional increase in Cmax and AUC from time 0 to 24 hours after dosing (AUC[0-24]) from 50 to 320 mg. The exposure on Day 14 was, on average, 1.9- to 2.3-fold higher than that of Day 1 for Cmax and 2.2- to 2.6-fold higher than Day 1 for AUC(0-24). Detailed summary statistics are available in the Study Synopsis [GSK Document Number 2018N375461 00].

#### 2.2.3. Preliminary Safety and Pharmacokinetic Data in Study 208131

The FTIH Study 207187 used a bis-hydrochloride salt capsule formulation of GSK3640254, which is not suitable for long-term clinical development.

Study 208131 was a single-center, open-label, 2-period, 2-sequence crossover design, conducted in 14 healthy participants in the United Kingdom. This study was designed to assess the relative BA of the formulation planned for Phase 2a (mesylate salt in a capsule) to the FTIH formulation (bis-hydrochloride salt in a capsule) administered following a moderate calorie and fat meal. All participants completed dosing and the blinded preliminary safety data showed a total of 11 AEs (all Grade 1). Two AEs of headache were related to study drug. The most common AE was headache (3 instances). There were 3 GI AEs (abdominal pain, bleeding gums, and flatulence). There were no cardiac or psychiatric AEs. There were no clinically significant changes in vital signs, ECG parameters, or safety laboratory parameters.

Preliminary PK results from Study 208131 showed that in the presence of a moderate fat meal, the relative BA of GSK3640254 following 200 mg GSK3640254 mesylate salt administration relative to 200 mg GSK3640254 bis-hydrochloride salt administration was 110% and 116% based on AUC from time zero extrapolated to infinity and Cmax, respectively.

#### 2.3. Benefit/Risk Assessment

Based upon preclinical and clinical studies, the major risks for GSK3640254 are GI intolerability (e.g., abdominal pain and diarrhea) and toxicity (e.g., single-cell parietal cell necrosis), prolongation of the QTc, and neuropsychiatric safety. Reproduction of preclinical GI toxicity findings would be unlikely during the limited dosing of GSK3640254 in this study. One preclinical study showed 1 dog with an increased QTc interval when given a single dose of GSK3640254. As described in Section 2.2.2, a cardiodynamic analysis of healthy participants in Study 207187 was conducted. A final model from the MAD data showed a QT effect (ΔΔQTcF) of GSK3640254 could be predicted to be 5.38 ms (90% CI: 1.66 to 9.10) and 6.70 ms (90% CI: 2.79 to 10.61) for the 200 mg (1779 ng/mL) and 320 mg (2154 ng/mL) doses, respectively, on Day 14. Based on this concentration-QTc analysis, a QTcF effect above 10 ms could be excluded up to GSK3640254 plasma concentrations of approximately 2000 ng/mL (corresponding to doses approximately ≤200 mg QD; note, 200 mg QD is the dose used in this study). Importantly, there were no abnormal clinically significant arrhythmias or QTc prolongations (values >500 ms or increases >60 ms from Baseline) in Study 207187. This study contains specific cardiac exclusion criteria, has ECG monitoring (at Tmax once GSK3640254 attains steady state concentration), and has QTcF-based stopping criteria.

Finally, the protocol will exclude potential participants with any significant pre-existing psychiatric condition or positive (abnormal) response confirmed by the investigator on a clinician (or qualified designee)-administered Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS assessment will also be administered by a clinician (or qualified designee) during the on-treatment portion of the study.

To ensure the overall safety of participants (including, but not limited to, the risk of GI intolerability, QTc prolongation, and neuropsychiatric safety), this clinical study will include healthy adults who will receive clinical, ECG, and laboratory evaluations during their participation. More detailed information about the known and expected benefits and risks and reasonably expected AEs of GSK3640254 may be found in the CIB [GSK Document Number 2018N379610 00).

2018N383392\_00 **CONFIDENTIAL** 209713

## 2.3.1. Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Investigational Product (IP) GSK3640254 | | |
| Cardiovascular (QT prolongation) | Preclinically, GSK3640254 inhibited cardiac hERG/IKr potassium, cardiac SCN5A sodium and L-type calcium channel currents recorded from HEK 293 cells stably transfected with complementary Deoxyribonucleic acid (DNA) from the ion channels. In a single-dose safety pharmacology study in telemeterized dogs, increases in QT interval (up to 20 ms) occurred primarily in 1 dog given 17 mg/kg. Later, there were no GSK3640254-related effects on ECG parameters in dogs given up to 25 mg/kg/day for 4 weeks. In the first time in human study 207187, no participant exhibited QTc change from Baseline >60 ms or QTc >500 ms. As described in Section 2.3, in the concentration-QTc analysis, a QTcF effect above 10 ms could be excluded up to GSK3640254 plasma concentrations of approximately 2000 ng/mL (corresponding to doses approximately ≤200 mg QD). | Screening: Protocol exclusion criteria based on Screening ECG parameters and cardiac medical history. On-Treatment: Participants will have ECG monitoring (at a clinically reasonable frequency) during the course of the study (see SoA, Section 1.3) with QTc stopping criteria (see Section 7.1.2). |
| GI intolerability and toxicity | Clinical signs indicative of GI intolerability (sporadic vomiting and abnormal feces beginning on Day 1 and continuing throughout the dosing periods) occurred mainly in dogs at ≥1 mg/kg/day. | Screening: Protocol exclusion criterion based on pre-existing GI pathology or Baseline GI signs/symptoms. |
| | Additionally, toxicity findings of single-cell necrosis | On-Treatment: Participants will undergo |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | of parietal cells and/or chief cells were present in preclinical species. These findings were reversible. Gastrointestinal intolerability (predominantly abdominal pain and diarrhea) was seen with a structurally related compound GSK3532795 which was evaluated through Phase 2b dosing. | continuous evaluation for AEs during their participation in the study; there will be individual clinical stopping criteria based upon intensity of treatment-emergent AEs. A GI toxicity evaluation and monitoring plan will be available to guide investigators should GI AEs emerge (see |
| | In the multiple ascending dose part of the first time in human study 207187, clinically relevant GI AEs (abdominal pain lower, diarrhoea, feces soft, gastro-esophageal reflux disease, nausea, abdominal distention, and abdominal pain) were experienced by 9 subjects. The greatest incidences were in the GSK3640254 200 mg arms (Cohorts 5 and 7) but ultimately, no dose/AE relationship was apparent. One subject each in the GSK3640254 200 mg arm and blinded 320 mg arm reported nausea (mild in intensity), considered by the investigator in each case to be related to study drug. | Section 8.2.6). |
| Neurologic/psychiatric safety | Two psychiatric SAEs in previous maturation inhibitor GSK3532795 clinical program (acute psychosis, homicidal/suicidal ideation) were seen at supratherapeutic doses in healthy participants in the thorough QT (TQT) study. From a neurologic and psychiatric AE summary and PK/pharmacodynamic analysis for | Screening: Protocol exclusion criterion based on any pre-existing psychiatric condition (including results of psychological assessment) for participants. Participants will have a clinician (or qualified designee) administered C-SSRS and will be included given no positive (abnormal) response. On-Treatment: Participants will undergo physical |
| | GSK3532795 across all studies Grade 1 headache and Grade 1 sleep abnormalities were the | examinations and laboratory testing. In addition, participants will undergo continuous evaluation for |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | predominant AEs, with a trend for increasing neurologic and psychiatric AEs with increasing dose (based on TQT and Phase 2b studies). No exposure-response relationship was seen for select neurologic and psychiatric AEs (based on TQT and Phase 2b studies). Central nervous system penetration data for GSK3532795 and GSK3640254 in rats demonstrate a similarly low brain distribution/penetration. In the multiple ascending dose part of first time in human study 207187, clinically relevant preferred terms from the system organ class nervous system were experienced by 5 subjects (somnolence, disturbance in attention, and lethargy) and showed that the greatest incidence arose in the GSK3640254 200 mg arms (Cohorts 5 and 7), but no dose/AE relationship was apparent. Seven subjects experienced five psychiatric AEs: agitation, abnormal dreams, insomnia, depressed mood, and nightmare. All events were mild in intensity and considered by the investigator to be unrelated to study drug, apart from one subject from the blinded 320 mg arm who experienced lethargy which was considered related to study drug | AEs during their participation in the study; there are individual clinical stopping criteria and monitoring based upon incidence and intensity of treatment-emergent psychiatric AEs (Section 7.1.4 and Section 8.2.5). Participants will be housed throughout study conduct to ensure rapid diagnosis and management of any potential event. The C-SSRS will be administered during and after the treatment phase of the study. In the event of a positive (abnormal) response confirmed by the investigator, the participant will discontinue from the trial and the investigator will arrange for urgent specialist psychiatric evaluation and management. Guidance for the investigator on the management of emergent psychiatric symptoms will be available. |

#### 2.3.2. Benefit Assessment

This is a study in healthy participants; no medical benefit will be derived by participants' participation.

#### 2.3.3. Overall Benefit: Risk Conclusion

Given the preclinical profile of GSK3640254, the clinical profile of a structurally similar MI (GSK3532795), the clinical data gathered from Studies 207187 and 208131, and the planned clinical procedures and evaluations in this study, the potential risks to participants receiving GSK3640254 are low, evaluable, and manageable.

#### 3. OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the relative bioavailability of<br>GSK3640254 mesylate tablets and<br>GSK3640254 mesylate capsules (in the<br>presence of a moderate fat meal) | <ul> <li>AUC(0-∞), AUC(0-t), Cmax, and Tmax for<br/>GSK3640254</li> </ul> |
| To assess the effect of food (fasted,<br>moderate fat meal, and high fat meal) on<br>the PK of the GSK3640254 mesylate tablet<br>formulation | |
| Secondary | |
| To assess the safety and tolerability of<br>GSK3640254 following single oral<br>administration to healthy participants under<br>fasted or fed (moderate fat or high fat)<br>conditions | <ul> <li>Safety and tolerability parameters for<br/>AEs/SAEs, observed and change from<br/>Baseline clinical laboratory assessments,<br/>ECGs, and vital sign measurements</li> </ul> |
| To characterize the PK of GSK3640254 | • tlag, t1/2, CL/F, and Vz/F for GSK3640254 |
| | GSK3640254 PK concentrations in plasma |

AE = adverse event;  $AUC(0-\infty)$  = area under the plasma concentration-time curve from time zero extrapolated to infinity; AUC(0-t) = area under the plasma concentration-time curve from time zero to time t; CL/F = apparent oral clearance; Cmax = maximum observed concentration; ECG = electrocardiogram; PK = pharmacokinetics; SAE = serious adverse event; t1/2 = apparent terminal phase half-life; tlag = lag time for absorption; Tmax = time of maximum observed concentration; Vz/F = apparent volume of distribution.

#### 4. STUDY DESIGN

# 4.1. Overall Design

This is a Phase 1, randomized, open-label, single-dose, 4-period crossover study to compare the relative BA of a tablet formulation of GSK3640254 with the capsule

formulation and to assess the effect of food on the PK of the tablet formulation in healthy participants.

The study will consist of a Screening period and 4 sequential treatment periods with a single dose of study intervention per treatment period. Prior to dosing on Day 1 of Period 1, participants will be randomly assigned to 1 of 4 treatment sequences (ABCD, BADC, CDAB, or DCBA). Participants will receive each of the following treatments administered as 1 treatment per period:

- Treatment A: GSK3640254 200 mg (single dose given as 2 × 100-mg capsules) administered under moderate fat conditions (reference).
- Treatment B: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under moderate fat conditions (test).
- Treatment C: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under fasted conditions (reference).
- Treatment D: GSK3640254 200 mg (single dose given as  $2 \times 100$ -mg tablets) administered under high fat conditions (test).

To ensure adequate washout, there will be at least 7 days between each dose of study intervention, with an allowance window of 4 hours (i.e., 7 days minus 4 hours) to allow flexibility in scheduling participants for dosing at the clinic. Treatments A, B, and D will be administered in the fed state. Participants will fast overnight for at least 10 hours prior to dosing and will receive a moderate fat (Treatments A and B) or high fat (Treatment D) meal 30 minutes prior to dosing. Dose administration will occur within 5 minutes of completion of meal consumption. Participants will not receive any further food until 4 hours after dosing. Treatment C will be administered in the fasted state. Participants will fast overnight for at least 10 hours prior to dosing and until 4 hours after dosing.

Pharmacokinetic blood samples for the analysis of GSK3640254 will be collected prior to dosing (0 hour) on Day 1 and up to 96 hours postdose in Periods 1, 2, 3, and 4.

Safety and tolerability will be assessed by monitoring and recording of AEs, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings.

Study assessments will be performed as indicated in the SoA (Section 1.3). Study participants will be confined to the clinic from Day –1 until discharge on Day 5 of Period 4. The total duration of the study, including Screening, is approximately 54 days.

# 4.2. Scientific Rationale for Study Design

This is an open-label, single-dose, 4-period crossover study to compare the relative BA of the GSK3640254 formulation planned for Phase 2b (mesylate salt in a tablet) with the Phase 2a formulation (mesylate salt in a capsule) when administered following a moderate calorie and fat meal. In addition, this study will investigate the effect of food on the PK of the GSK3640254 mesylate tablet formulation.

The effect of food on the PK of a structurally similar HIV-1 MI (GSK3532795) was previously evaluated: AUC increased 1.8-, 2.1-, and 2.5-fold when a single dose of 180 mg GSK3532795 was given with a light, moderate, or high fat meal, respectively, as compared to administration under fasting conditions [GSK Document Number 2017N322200\_00]. All GSK3640254 clinical studies to date, including a Phase 2a proof of concept study, have been conducted with moderate calorie and fat meals. It is intended that this will be the only food-effect BA clinical study for GSK3640254; therefore, this study will investigate the effect of moderate and high calorie and fat meals on the PK, safety, and tolerability of the GSK3640254 mesylate tablet formulation, as compared to administration under fasting conditions.

The open-label crossover design of this study is well-established for evaluation of the relative BA of different oral dosage forms and for studying the effect of food on BA. Random assignment to treatment sequences is an attempt to prevent bias. The washout of at least 7 days between each dose of study intervention should eliminate the possibility of carryover of drug exposure from the previous dose. There are appropriately named "test" and "reference" study treatments, which will be evaluated for the relative BA comparisons.

This study is participant to the appropriate regulatory and ethics committee approval and will be listed on the website ClinicalTrials.gov. No blinding or placebo control will be used, as these are not necessary for the purposes of this study.

#### 4.3. Justification for Dose

The dose of 200 mg GSK3640254 was selected for this study as the maximum projected clinically therapeutic dose of GSK3640254 is 200 mg QD. The t1/2 of GSK3640254 was approximately 22 hours in the MAD portion of Study 207187 at the 200-mg dose. To ensure adequate washout, there will be at least 7 days between each dose of study intervention, with an allowance window of 4 hours (i.e., 7 days minus 4 hours) to allow flexibility in scheduling participants for dosing at the clinic.

## 4.4. End-of-Study Definition

A participant is considered to have completed the study if he or she has completed all phases of the study including the final date on which data were or are expected to be collected.

The end of the study is defined as the date of the last visit of the last participant in the study or last scheduled procedure shown in the SoA (Section 1.3) for the last participant in the study.

#### 5. STUDY POPULATION

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all the following criteria apply:

#### Age

1. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.

#### Type of Participant and Disease Characteristics

2. Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).

#### Weight

3. Body weight  $\geq$ 50.0 kg (110 lbs) for men and  $\geq$ 45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kg/m<sup>2</sup> (inclusive).

#### Sex

Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

- 4. Male or female
  - a. Female participants:
    - 1. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:
      - Is not a woman of childbearing potential (WOCBP) as defined in Appendix 3.

#### OR

- Is a WOCBP and using a nonhormonal contraceptive method that is highly effective, with a failure rate of <1%, as described in Appendix 3 for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
- 2. A WOCBP must have a negative highly sensitive serum pregnancy test (Appendix 2) at Screening and Day –1.
- 3. Additional requirements for pregnancy testing during and after study intervention are outlined in Appendix 2.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

#### **Informed Consent**

5. Capable of giving signed informed consent as described in Appendix 4, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

#### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical History**

- 1. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
- 2. A pre-existing condition interfering with normal GI anatomy or motility (e.g., gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
- 3. Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
- 4. Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the VH/GSK Medical Monitor.
- 5. Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
- 6. Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.

#### **Laboratory Assessments**

- 7. Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
- 8. Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention AND positive on reflex to hepatitis C ribonucleic acid (RNA).
- 9. Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.

- 10. ALT >1.5 × upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
- 11. Bilirubin  $>1.5 \times$  ULN (isolated bilirubin  $>1.5 \times$  ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
- 12. Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
- 13. Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
- 14. A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.

#### **Prior/Concomitant Therapy**

- 15. Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study. (Note: acetaminophen/paracetamol at doses of ≤2 grams/day and topical hydrocortisone cream 1% are permitted for use any time during the study.)
- 16. Treatment with any vaccine within 30 days prior to receiving study intervention.
- 17. Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.

#### **Prior/Concurrent Clinical Study Experience**

- 18. Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
- 19. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.

#### **Diagnostic Assessments**

20. Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered C-SSRS.

- 21. Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, second-degree atrioventricular block Mobitz Type II, third-degree atrioventricular block, complete heart block, or conduction abnormality) which, in the opinion of the investigator or VH/GSK Medical Monitor, will interfere with the safety for the individual participant.
- 22. Exclusion criteria for Screening ECG (a single repeat is allowed for eligibility determination):

| | Males | Females |
|---|---|---|
| Heart rate 1 | <45 or >100 bpm | <50 or >100 bpm |
| QTcF interval <sup>2</sup> (Fridericia's) | >450 ms | >450 ms |

A heart rate from 100 to 110 bpm can be rechecked by electrocardiogram or vital signs within 30 minutes to verify eliqibility.

#### **Other Exclusions**

- 23. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
- 24. Unable to refrain from tobacco or nicotine-containing products within 3 months prior to Screening.
- 25. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

## 5.3. Lifestyle Considerations

# 5.3.1. Meals and Dietary Restrictions

- Refrain from excessive consumption of red wine, grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study. Excessive consumption is defined as more than one glass of wine or juice or one of these fruits per day, in combination.
- Treatments A, B, and D will be administered in the fed state. The participants will fast overnight for at least 10 hours prior to dosing and will receive a moderate fat (Treatments A and B) or high fat (Treatment D) meal 30 minutes prior to dosing. Participants will eat this meal in 30 minutes or less. Dose administration will occur within 5 minutes of completion of meal consumption. Participants will not receive any further food until 4 hours after dosing on serial PK sampling days (e.g., Day 1 of Periods 1, 2, 3, and 4). The moderate fat meal will contain about 600 calories with approximately 30% of the calories coming

<sup>2</sup> The QTc is the QT interval corrected for heart rate using Fridericia's formula (QTcF). It is either machine read or manually over-read. The specific formula used to determine eligibility and discontinuation for an individual participant will be Fridericia's formula.

from fat. The high fat meal will contain about 800 to 1000 calories with approximately 50% of the calories coming from fat (DHHS, 2002).

- Treatment C will be administered in the fasted state. The participants will fast overnight for at least 10 hours prior to dosing until 4 hours after dosing.
- No water is allowed from 1 hour prior to dosing until 1 hour after dosing except for the glass of water needed to administer the study intervention (e.g., 240 mL).
   Water is allowed ad libitum at all other times.
- A standard lunch will be provided 4 hours after dosing. A standard dinner will be served approximately 10 hours after dosing. The food content of meals must be identical on serial PK sampling days (e.g., Day 1 of Periods 1, 2, 3, and 4).

### 5.3.2. Caffeine, Alcohol, and Tobacco

- Participants will abstain from ingesting caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) for 24 hours before the start of dosing until after collection of the final PK sample.
- Participants will abstain from alcohol for 48 hours before the start of dosing until after collection of the final PK sample.
- Use of tobacco and nicotine-containing products will not be allowed from 3 months prior to Screening until after the final visit.
- Participants must have a negative drug test at Screening and Day –1 and must abstain from recreational drug use from Screening until after the final visit.

#### 5.3.3. Activity

• Participants will abstain from strenuous exercise for 24 hours before each blood collection for clinical laboratory tests. Participants may participate in light recreational activities during studies (e.g., watching television, reading).

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAEs.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be rescreened.

#### 6. STUDY INTERVENTION

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

6.1. Study Interventions Administered

| Intervention Name | GSK3640254 | GSK3640254 |
|---|---|---|
| Туре | drug | drug |
| Dose Formulation | tablet | capsule |
| Unit Dose Strength(s) | 100 mg | 100 mg |
| Dosage Level(s) | 200 mg, single dose | 200 mg, single dose |
| Route of Administration | oral | oral |
| IMP and NIMP | IMP | IMP |
| Sourcing | Provided centrally by the Sponsor | Provided centrally by the Sponsor |
| Packaging and<br>Labeling | Provided in high-density polyethylene bottles. Each bottle will be labelled as required per country requirement. | Provided in high-density polyethylene bottles. Each bottle will be labelled as required per country requirement. |

IMP = investigational medicinal product; NIMP = non-investigational medicinal product

# 6.2. Preparation/Handling/Storage/Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study interventions must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.
- 3. The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).
- 4. Further guidance and information for the final disposition of unused study intervention are provided in the Study Reference Manual (SRM).
- 5. Under normal conditions of handling and administration, study intervention is not expected to pose significant safety risks to site staff.
- 6. A Material Safety Data Sheet/equivalent document describing occupational hazards and recommended handling precautions either will be provided to the investigator, where this is required by local laws, or is available upon request from VH/GSK.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

This is an open-label study. Study participants will be randomly assigned to 1 of 4 treatment sequences (ABCD, BADC, CDAB, or DCBA) in accordance with the randomization schedule generated by PPD prior to the start of the study and using validated software.

## 6.4. Study Intervention Compliance

- When the individual dose for a participant is prepared from a bulk supply, the preparation of the dose will be confirmed by a second member of the study site staff.
- When participants are dosed at the site, they will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of each dose administered in the clinic will be recorded in the source documents. The dose of study intervention and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention. Study site personnel will examine each participant's mouth to ensure that the study intervention was ingested.

## 6.5. Concomitant Therapy

Acetaminophen/paracetamol at doses of ≤2 grams/day and topical hydrocortisone cream 1% are permitted for use any time during the study and their use should be documented in the case report form (CRF). Other medications are not permitted without prior discussion with the VH/GSK medical monitor.

#### 6.6. Dose Modification

Not applicable.

# 6.7. Intervention After the End of the Study

Participants will not receive any additional treatment from VH/GSK, or with GSK3640254, after the completion of the study because only healthy participants are eligible for study participation.

# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 7.1. Discontinuation of Study Intervention

In rare instances, it may be necessary for a participant to permanently discontinue study intervention. If study intervention is permanently discontinued, the participant will remain in the study to be evaluated for safety. See the SoA (Section 1.3) for data to be collected at the time of discontinuation of study intervention.

#### 7.1.1. Liver Chemistry Stopping Criteria

Liver chemistry stopping and increased monitoring criteria have been designed to assure participant safety and evaluate liver event etiology (in alignment with the Food and Drug Administration premarketing clinical liver safety guidance:

https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM174090.pdf).

Discontinuation of study intervention for abnormal liver tests is required when a participant has an ALT  $\geq$ 3 × ULN or if the investigator believes study intervention discontinuation is in the best interest of the participant.

Details of liver safety follow-up procedures are described in Appendix 5.

# 7.1.1.1. Study Intervention Restart or Rechallenge After Liver Stopping Criteria Met

Study intervention restart or rechallenge after liver chemistry stopping criteria are met by any participant in this study is not allowed.

## 7.1.2. QTc Stopping Criteria

The *same* correction formula (QTcF) *must* be used for *each individual participant* to determine eligibility for and discontinuation from the study. This formula may not be changed or substituted once the participant has been enrolled.

- The Baseline QTcF should be based on averaged QTcF values of triplicate ECGs obtained over a brief (e.g., 5-10 minute) recording period from the Day -1 ECG.
- A randomized participant that develops an on-treatment QTcF >500 ms or an increase from Baseline QTcF >60 ms should have two repeat unscheduled ECGs within 10 minutes. Using these triplicate ECGs, if the average QTcF >500 ms or an increase from Baseline QTcF >60 ms, the participant will be withdrawn from the study. Finally, this participant should have repeated unscheduled ECGs until their QTcF measurement returns to their original averaged QTcF value at Day -1.

See the SoA (Section 1.3) for data to be collected at the time of treatment discontinuation and follow-up and for any further evaluations that need to be completed.

#### 7.1.3. Columbia Suicide Severity Rating Scale Criteria

Emergence of any positive (abnormal) response confirmed by the investigator on a clinician (or qualified designee) administered C-SSRS during the treatment phase of the study will be cause for discontinuation of study intervention.

Refer to the SoA (Section 1.3) for data to be collected at the time of intervention discontinuation and follow-up and for any further evaluations that need to be completed.

# 7.1.4. Individual Participant Laboratory Abnormality and Adverse Event Stopping Criteria

Investigators should make every effort to have a discussion with the medical monitor before the next dose to help assess if the study intervention should be stopped.

- Any clinically significant AE deemed to require discontinuation of study intervention
- Any Grade 3 or higher rash or Grade 2 rash with evidence of systemic involvement
- Any allergic or hypersensitivity reactions to either or both drugs
- Any Grade 3 or higher psychiatric AE
- New onset suicidal ideation
- Any Grade 3 or higher AE related to study intervention
- Any Grade 4 AE or laboratory abnormalities (with the exception of an asymptomatic Grade 4 cholesterol, triglyceride, or CPK increase)

## 7.2. Participant Discontinuation/Withdrawal From the Study

- A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance or administrative reasons. This is expected to be uncommon.
- A participant who is withdrawn from the study for any reason related to safety (listed in Section 7.1.4 or otherwise) will be continued to be followed to assess the outcome of the safety event that triggered discontinuation of study intervention.
- At the time of discontinuing from the study, if possible, an early discontinuation visit should be conducted, as shown in the SoA. See SoA (Section 1.3) for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.
- The participant will be permanently discontinued both from the study intervention and from the study at that time.
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.

## 7.3. Lost to Follow-Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

Discontinuation of specific sites or of the study as a whole are handled as part of Appendix 4.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and their timing are summarized in the SoA (Section 1.3).
- Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All Screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a Screening log to record details of all participants screened and to confirm eligibility or record reasons for Screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (e.g., blood count) and obtained before signing of ICF may be utilized for Screening or Baseline purposes provided the procedure met the protocol-specified criteria and was performed within the time frame defined in the SoA.
- The maximum amount of blood collected from each participant over the duration of the study, including any extra assessments that may be required, will not exceed 500 mL.

• Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

# 8.1. Efficacy Assessments

Not applicable.

## 8.2. Safety Assessments

Planned time points for all safety assessments are provided in the SoA (Section 1.3).

## 8.2.1. Physical Examinations

- A full physical examination will include, at a minimum, assessments of the skin, cardiovascular, respiratory, GI, and neurological systems. Height and weight will also be measured and recorded.
- A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
- Investigators should pay special attention to clinical signs related to previous serious illnesses.

### 8.2.2. Vital Signs

- Oral temperature, pulse rate, respiratory rate, and blood pressure will be assessed.
- Blood pressure and pulse measurements will be assessed in the semi-recumbent position with a completely automated device. Manual techniques will be used only if an automated device is not available.
- Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones).
- At each time point at which triplicate measurements are required, 3 consecutive blood pressure and pulse readings will be recorded at intervals of at least 1 minute. Each measurement will be recorded in the CRF.
- When vital signs are scheduled at the same time as blood collections for laboratory tests, vital signs are to be taken first.

#### 8.2.3. Electrocardiograms

- Twelve-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals. Refer to Section 7.1.2 for QTcF withdrawal criteria and additional QTcF readings that may be necessary.
- Twelve-lead ECGs will be performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes.

At each time point at which triplicate ECGs are required, 3 individual ECG tracings should be obtained as closely as possible in succession, but no more than 2 minutes apart. The full set of triplicates should be completed over a brief (e.g., 5 to 10 minutes) recording period. Each measurement will be recorded in the CRF.

#### 8.2.4. Clinical Safety Laboratory Assessments

- Refer to Appendix 2 for the list of clinical laboratory tests to be performed.
- The investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF. The laboratory reports must be filed with the source documents. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- All laboratory tests with values considered clinically significantly abnormal during participation in the study or within 7 days after the last dose of study intervention should be repeated until the values return to normal or Baseline or are no longer considered significantly abnormal by the investigator or medical monitor.
- If such values do not return to normal/Baseline within a period of time judged reasonable by the investigator, the etiology should be identified, and the sponsor notified.
- All protocol-required laboratory assessments, as defined in Appendix 2, must be conducted in accordance with the laboratory manual and the SoA.

# 8.2.5. Suicidal Risk Monitoring and Management of Emergent Psychiatric Symptoms

GSK3640254 is not a central nervous system active drug nor is it being developed for a neurologic or psychiatric condition. However, given the risk of suicidal ideation identified with previous MI GSK3532795, all participants will undergo Screening using the C-SSRS administered by a clinician (or qualified designee); any positive (abnormal) response confirmed by the investigator, will exclude them from participating. A repeat assessment will be done during the treatment phase of the study. In case of positive (abnormal) response confirmed by the investigator, the participant will discontinue from the trial and the investigator will arrange for urgent specialist psychiatric evaluation and management.

As described in Section 7.1.4, new onset suicidal ideation at any time will result in immediate discontinuation from the trial and the investigator will arrange for urgent specialist psychiatric evaluation and management.

The definitions of behavioral suicidal events used in this scale are based on those used in the Columbia Suicide History Form [Posner, 2007]. Questions are asked on suicidal behavior, suicidal ideation, and intensity of ideation. Screening visit questions will be in

relation to lifetime experiences and current experiences (within the past 2 months) and all subsequent questioning in relation to the last assessment.

Emergent non-suicidal psychiatric AE evaluation and management:

- Any Grade 1 or 2 psychiatric AE: A Grade 1 or 2 psychiatric AE may result in
  additional unscheduled visits (in-clinic or at home) as clinically indicated. This
  may include a more in-depth assessment of AE through interview, additional
  unscheduled clinical labs, and/or imaging. Psychiatric consultation may be
  required at the discretion of the investigator. Any pharmacotherapy should be
  discussed with the medical monitor.
- Any Grade 3 or 4 psychiatric AE: As described in Section 7.1.4, a Grade 3 or 4 psychiatric AE will result in discontinuation from the trial and emergency psychiatric evaluation (including potential hospitalization and pharmacotherapy as indicated).

## 8.2.6. Gastrointestinal Toxicity Evaluation and Monitoring Plan

Preclinical toxicology studies in rats and dogs have suggested a potential for GI-related toxicity with GSK3640254. This section provides general guidance to the investigator on the evaluation and management of primarily upper GI symptoms (Table 1). The investigator may contact the VH/GSK Medical Monitor to discuss evaluation and management (including discontinuation of a participant) of any GI symptoms throughout the study.

Table 1 Gastrointestinal Toxicity Evaluation and Management

| HISTORY | For symptoms of all grades, a thorough history forms the foundation of proper evaluation and management. The following are potential manifestations of some GI clinical syndromes that may occur (possibly in combination) during the clinical study. |
|---|---|
| Nausea and Vomiting | The investigator should attempt to identify the etiology of these symptoms (and whether it is intraperitoneal, extraperitoneal, medication related, infection related, or due to a metabolic disorder (Hasler, 2012). Medications can cause nausea and vomiting acutely. |
| Dyspepsia | The investigator should identify the presence of red flags (odynophagia, unexplained weight loss, recurrent vomiting, GI bleeding, jaundice, palpable mass or adenopathy, or family history of GI malignancy). Symptoms of dyspepsia could include early satiety, bloating, or belching. Additionally, atypical symptoms of dyspepsia could include: pharyngitis, asthma, bronchitis, hoarseness, chest pain, or abdominal pain. |
| Other Clinical<br>Syndromes | Additional diagnostic criteria for other GI disorders potentially encountered in the clinical study are available elsewhere (Rome Foundation, 2019). |

| PHYSICAL<br>EXAMINATION | Physical examination should complement elements obtained from the history (Hasler, 2012). Acutely, the investigator may assess for signs of intravascular volume depletion (e.g., orthostasis) and/or aspiration of vomitus as appropriate. Abdominal tenderness and guarding may indicate inflammation. The presence of fecal blood can indicate mucosal damage (e.g., from an ulcer). Complete evaluation of dyspepsia should include an oral examination (poor dentition or pharyngeal erythema) and lungs for wheezing. |
|---|---|
| DIAGNOSTIC<br>EVALUATION AND<br>MANAGEMENT | A major goal in the diagnostic evaluation of a participant with upper GI symptoms is to quickly arrive at a final diagnosis without exposing the participant to unnecessary (invasive) testing; investigators should exercise good clinical judgment in this regard (Soll, 2009). A major goal of therapy is directed at correcting the underlying identifiable medical or surgical abnormalities. Consultation (e.g., gastroenterologist) is recommended as clinically indicated. |
| Grade 1 symptoms | Participants may be treated symptomatically. If participants develop dyspepsia alone, generally only limited and direct diagnostic testing should be performed. If the participant has dyspepsia they should limit alcohol, caffeine, chocolate, tobacco, and eating directly before bedtime. |
| Grade 2 symptoms | <ul> <li>Diagnostic testing may include but is not limited to the following (as clinically indicated):</li> <li>Serum chemistries and assessment of hemoglobin if not recently performed</li> <li>Testing for <i>Helicobacter pylori</i></li> <li>Polymerase chain reaction for viruses (e.g., cytomegalovirus)</li> <li>For participants who are infected with <i>H. pylori</i>, discontinuation from the study is necessary. Management should be targeted at addressing the underlying pathology.</li> </ul> |
| Grade 3 symptoms <sup>1</sup> | Diagnostic testing may include but is not limited to the following (as clinically indicated): The testing outlined above in Grade 2 A barium swallow Computed tomography scan to identify GI inflammation Upper endoscopy with biopsy as indicated (e.g., mucosal injury or the presence of red flags) Management should be targeted at addressing the underlying pathology. |
| Grade 4 symptoms 1 | Diagnostic testing may include but is not limited to the following (as clinically indicated): • The testing outlined above in Grade 2 and Grade 3 • An acute abdominal series Initial management can include correction of hemodynamic and electrolyte abnormalities as clinically indicated. After stabilization, management should be targeted at addressing the underlying pathology. |

GI = gastrointestinal.

A Grade 4 or related Grade 3 AE: The Investigator will discontinue the participant from the study and perform an evaluation/management plan incorporating element above.
#### 8.3. Adverse Events and Serious Adverse Events

The definitions of an AE or SAE can be found in Appendix 6. As described in Appendix 6, intensity of AEs (and laboratory abnormalities) will be graded using the most recent version of the Division of AIDS (DAIDS) grading table at the time of the last participant last visit. While the study population will consist of HIV-1 seronegative healthy participants, the DAIDS criteria will be used in later phase clinical studies (Phase 2a and beyond); additionally, the DAIDS criteria have a more conservative grading scale relative to other scales (e.g., Common Terminology Criteria for Adverse Events [CTCAE] v 4.0). Thus, participant safety evaluation and monitoring will be more conservative.

The investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE, and remain responsible for following up AEs that are serious, considered related to the study intervention or the study, or that caused the participant to discontinue the study (see Section 7).

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

- All SAEs will be collected from the signing of the ICF until the end of the study at the time points specified in the SoA (Section 1.3).
- All AEs will be collected from the start of intervention until the end of the study at the time points specified in the SoA (Section 1.3).
- Medical occurrences that begin before the start of study intervention but after obtaining informed consent will be considered medical history, not an AE, and will be recorded in the source documents.
- All SAEs will be recorded and reported to the sponsor or designee immediately
  and under no circumstance should this exceed 24 hours, as indicated in
  Appendix 6. The investigator will submit any updated SAE data to the sponsor
  within 24 hours of it being available.
- Investigators are not obligated to actively seek AEs or SAEs after the conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

## 8.3.2. Method of Detecting AEs and SAEs

- The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 6.
- Care will be taken not to introduce bias when detecting AE and/or SAE. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

#### 8.3.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs will be followed until the event is resolved, stabilized, otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3). Further information on follow-up procedures is given in Appendix 6.

## 8.3.4. Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the sponsor of a SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, Institutional Review Board (IRB) / Independent Ethics Committee (IEC), and investigators.
- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSARs) according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing a SAE or other specific safety information (e.g., summary or listing of SAEs) from the sponsor will review and then file it along with the CIB and will notify the IRB/IEC, if appropriate according to local requirements.

## 8.3.5. Pregnancy

- Details of all pregnancies in female participants will be collected after the start of study intervention and through the end of pregnancy (termination or delivery).
- If a pregnancy is reported, the investigator should inform VH/GSK within 24 hours of learning of the pregnancy.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.

#### 8.4. Treatment of Overdose

For this study, any dose of GSK3640254 greater than the planned dose within a 24-hour time period (±2 hours) will be considered an overdose.

VH/GSK does not recommend specific treatment for an overdose. The investigator will use clinical judgment to treat an overdose.

In the event of an overdose, the investigator should:

- 1. Contact the medical monitor immediately.
- 2. Closely monitor the participant for AE/SAE and laboratory abnormalities until GSK3640254 can no longer be detected systemically (at least 5 days).
- 3. Obtain a plasma sample for PK analysis immediately and through 7 days after the date of the last dose of study intervention if requested by the medical monitor (determined on a case-by-case basis).
- 4. Document the quantity of the excess dose as well as the duration of the overdosing in the CRF.

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the medical monitor based on the clinical evaluation of the participant.

#### 8.5. Pharmacokinetics

- Whole blood samples of approximately 2 mL will be collected for measurement of plasma concentrations of GSK3640254 as specified in the SoA (Section 1.3).
- A maximum of 10 samples may be collected at additional time points during the study if warranted and agreed upon between the investigator and the sponsor. Instructions for the collection and handling of biological samples will be provided by the sponsor. The actual date and time (24-hour clock time) of each sample will be recorded.
- Samples will be used to evaluate the PK of GSK3640254. Samples collected for analyses of GSK3640254 plasma concentration may also be used to evaluate safety aspects related to concerns arising during or after the study.
- Once the plasma has been analyzed for GSK3640254, any remaining plasma may be analyzed for other compound-related metabolites and the results reported under a separate protocol.

## 8.6. Pharmacodynamics

Not applicable.

#### 8.7. Genetics

A 6-mL blood sample for DNA isolation will be collected from participants who have consented to participate in the genetics analysis component of the study. Participation is optional. Participants who do not wish to participate in the genetic research may still participate in the study.

In the event of DNA extraction failure, a replacement genetic blood sample may be requested from the participant. Signed informed consent will be required to obtain a replacement sample unless it was included in the original consent.

See Appendix 7 for information regarding genetic research. Details on processes for collection and shipment and destruction of these samples can be found in the SRM.

#### 8.8. Biomarkers

Not applicable.

#### 8.9. Medical Resource Utilization and Health Economics

Medical Resource Utilization and Health Economics parameters are not evaluated in this study.

## 9. STATISTICAL CONSIDERATIONS

## 9.1. Statistical Hypotheses

There is no formal hypothesis that will be statistically tested in this study.

## 9.2. Sample Size Determination

## 9.2.1. Sample Size Assumptions

Based on the results from previous PK studies for GSK3640254 (GSK Study 207187 and 208131) the intra-subject coefficient of variability (CVw) ranged from 17%-38% and 13%-31%, respectively for AUC from time 0 to the end of the dosing interval (AUC $_{0-\tau}$ ) and Cmax. For recent PK study GSK 209712 the CVw were 7.8% and 11.5%, respectively for AUC $_{0-\tau}$ ) and Cmax. Therefore, it is decided that 38% would be a conservative estimate on which the sample size calculation is based.

Administration of GSK3640254 mesylate salt tablet formulation may change the exposure to GSK3640254 from the capsule formulation; therefore, a range for point estimate of 0.9, 1.0, and 1.1 were explored.

Administration of GSK3640254 with a high-fat meal compared to fasting is expected to increase the exposure to GSK3640254; therefore, a range for point estimate of 1.0, 1.1, and 1.2 were explored.

For GSK3640254, with a sample size of 12 evaluable participants, it is estimated that the precision (i.e. half-width of the 90% CI on the log and ratio scale), and CI on the original scale for each point estimate will be:

| Comparison | CVw<br>(%) | Half-Width<br>(log scale) | Half-Width<br>(original<br>scale) | Point<br>Estimate | 90% CI |
|---|---|---|---|---|---|
| GSK3640254 | | | | 0.9 | (0.688, 1.178) |
| | 0.309 | 1.0 | (0.764, 1.309) | | |
| | | | 1.1 | (0.841, 1.440) | |

209713

| Comparison | CVw<br>(%) | Half-Width<br>(log scale) | Half-Width<br>(original<br>scale) | Point<br>Estimate | 90% CI |
|---|---|---|---|---|---|
| GSK3640254 | <3640254 | | 1.0 | (0.764, 1.309) | |
| high fat meal to fasting | 38 | 0.269 | 0.309 | 1.1 | (0.841, 1.440) |
| | | | | 1.2 | (0.917, 1.570) |

## 9.2.2. Sample Size Sensitivity

For a sensitivity analysis, assuming a range of within-participant variability, a sample size of 12 evaluable participants, it is estimated that the precision (i.e. half-width of the 90% CI on the log and ratio scale), and CI on the original scale for each point estimate will be:

| Comparison | CVw (%) | Half-Width<br>(log scale) | Half-Width (original scale) | Point<br>Estimate | 90% CI |
|---|---|---|---|---|---|
| | | 0.073 | 0.076 | 0.9 | (0.837, 0.968) |
| | 10 | | | 1.0 | (0.930, 1.076) |
| | 10 | | | 1.1 | (1.023, 1.183) |
| | | | | 1.2 | (1.116, 1.291) |
| | | | | 0.9 | (0.779, 1.040) |
| Tablet to | 20 | 0.145 | 0.156 | 1.0 | (0.865, 1.156) |
| capsule | | | | 1.1 | (0.952, 1.272) |
| or | | | | 1.2 | (1.038, 1.387) |
| OI | | 0.215 0.240 | 0.9 | (0.726, 1.116) | |
| high fat meal | 30 | | 0.240 | 1.0 | (0.807, 1.240) |
| to fasting | | | | 1.1 | (0.887, 1.364) |
| | | | | 1.2 | (0.968, 1.488) |
| | 40 | 0.283 | 0.327 | 0.9 | (0.678, 1.194) |
| | | | | 1.0 | (0.754, 1.327) |
| | | | | 1.1 | (0.829, 1.460) |
| | | | | 1.2 | (0.904, 1.593) |

Approximately 16 participants (4 per treatment sequence) will be treated to ensure that 12 evaluable participants complete the study. If participants prematurely discontinue the

209713

study, additional participants may be randomized after consultation with the sponsor to ensure that 12 evaluable participants complete the study.

## 9.3. Populations for Analyses

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Screened | All participants who sign the ICF. |
| Safety | All participants who receive at least 1 dose of study medication. This population will be used for all demographic and safety summaries. |
| Pharmacokinetic Concentration | The PK Concentration Population will include all participants who undergo plasma PK sampling and have evaluable PK assay results. This population will be used for the PK concentration listings, summary tables, and plotting of concentration-time data. |
| Pharmacokinetic Parameter | The PK Parameter Population will include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated. This population will be used for PK parameter listings, summary tables, and statistical analysis tables. |

## 9.4. Statistical Analyses

## 9.4.1. Pharmacokinetic Analyses

Plasma GSK3640254 concentration-time data will be analyzed by PPD, under the oversight of Clinical Pharmacology Modeling & Simulation department within GSK, using noncompartmental methods with Phoenix WinNonlin Version 6.4 or higher. Statistical analysis will be performed by PPD, under the oversight of Clinical Statistics, GSK. Calculations will be based on the actual sampling times recorded during the study.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | The primary endpoints of this study are PK-related. The analysis for the primary PK endpoints will be performed for the PK Parameter Population. Plasma concentrations of GSK3640254 will be subjected to PK analyses using noncompartmental methods. |
| | <ul> <li>Based on the individual concentration-time data the following primary plasma PK parameters will be estimated:</li> <li>AUC(0-∞), AUC(0-t), Cmax, and Tmax</li> </ul> |

| Endpoint | Statistical Analysis Methods |
|---|---|
| | <ul> <li>Analysis will be performed to compare the relative BA of a tablet formulation of GSK3640254 with the capsule formulation, as appropriate. Analyses will be performed on the natural logarithms of AUC(0-∞), AUC(0-t), and Cmax using linear mixed-effect models with treatment, period, and sequence as fixed effects and participant as a random effect. Effects will be estimated, and CIs will be constructed for the following treatment comparison:</li> </ul> |
| | Treatment B (test) versus Treatment A (reference) |
| | Point estimates and 90% CIs for treatment differences on the log scale derived from the model will be exponentiated to obtain estimates for geometric mean ratios and CIs on the original scale. |
| | The effect of food (moderate or high fat meal) on the PK of the tablet formulation of GSK3640254 will be similarly analyzed for the following treatment comparisons: |
| | Treatment B (test) versus Treatment C (reference) |
| | Treatment D (test) versus Treatment C (reference) |
| | Non-parametric analysis will be performed to compare the Tmax of a tablet formulation of GSK3640254 with the capsule formulation, as appropriate. The Hodges-Lehmann estimate will be used to produce the median, median difference, and 90% CIs for the following comparison: |
| | Treatment B (test) versus Treatment A (reference) |
| | A p-value will be generated by the Wilcoxon signed-rank test |
| | The effect of food (moderate or high fat meal) on the Tmax of the tablet formulation of GSK3640254 will be similarly analyzed for the following comparisons: |
| | Treatment B (test) versus Treatment C (reference) |
| | Treatment D (test) versus Treatment C (reference) |
| | Summary statistics (arithmetic mean, geometric mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma GSK3640254 primary PK parameter values will be summarized by treatment. |
| Secondary | Based on the individual concentration-actual time data the following secondary plasma PK parameters will be estimated: |
| | • tlag, t1/2, CL/F, and Vz/F |
| | Summary statistics (arithmetic mean, geometric mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma GSK3640254 secondary PK parameter values will be summarized by treatment. |

| Endpoint | Statistical Analysis Methods |
|---|---|
| | Summary statistics (arithmetic mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma GSK3640254 PK concentrations will be summarized by treatment using the PK Concentration Population. |

## 9.4.2. Safety Analyses

All safety analyses will be performed on the Safety Population.

Safety data will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. No formal statistical analysis of the safety data will be conducted.

The details of the statistical analyses of safety data will be provided in the reporting and analysis plan.

#### 9.4.3. Other Analyses

Not applicable.

## 9.5. Interim Analyses

No interim analysis is planned.

## 9.5.1. Data Monitoring Committee (DMC)

Not applicable.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

## 10.1. Appendix 1: Abbreviations and Trademarks

| AE | Adverse event |
|---|---|
| ALT | Alanine aminotransferase |
| AUC | Area under the plasma concentration-time curve |
| AUC(0-24) | Area under the plasma concentration-time curve from time 0 to 24 hours after dosing |
| AUC(0-∞) | Area under the plasma concentration-time curve from time zero extrapolated to infinity |
| AUC(0-t) | Area under the plasma concentration-time curve from time zero to time t |
| AUC(0-τ) | AUC from time 0 to the end of the dosing interval |
| AST | Aspartate transaminase |
| BA | Bioavailability |
| BMS | Bristol-Myers Squibb |
| bpm | Beats per minute |
| CL/F | Apparent oral clearance |
| CI | Confidence interval |
| CIB | Clinical Investigator's Brochure |
| Cmax | Maximum observed concentration |
| CONSORT | Consolidated Standards of Reporting Trials |
| СРК | Creatine phosphokinase |
| CRF | Case report form |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CVw | Intra-subject coefficient of variability |
| DAIDS | Division of AIDS |
| DNA | Deoxyribonucleic acid |
| ECG | Electrocardiogram |
| FSH | Follicle-stimulating hormone |
| FTIH | First time in human |
| g | Grams |

| GCP | Good Clinical Practice |
|-------------------|-----------------------------------------------------|
| Gl | Gastrointestinal |
| GSK | GlaxoSmithKline |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human immunodeficiency virus |
| HRT | Hormonal replacement therapy |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| IDSL | Integrated Data Standards Library |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal product |
| INR | International normalized ratio |
| IP | Investigational product |
| IU/L | International units per liter |
| IRB | Institutional Review Board |
| kg | Kilograms |
| kg/m <sup>2</sup> | Kilograms per square meter |
| lbs | Pounds |
| MAD | Multiple-ascending dose |
| mg | Milligrams |
| mg/kg/day | Milligrams per kilogram per day |
| MI | Maturation inhibitor |
| mL | Milliliter |
| mm | Millimeter |
| ms | Milliseconds |
| ng/mL | Nanograms per milliliter |
| NIMP | Non-investigational medicinal product |
| PK | Pharmacokinetic(s) |
| QD | Once daily |
| QTc | Corrected QT interval |
| QTcF | Corrected QT interval using the Fridericia formula |
| RNA | Ribonucleic acid |

209713

| SAD | Single-ascending dose |
|-------|------------------------------------------------|
| SAE | Serious adverse event |
| SoA | Schedule of activities |
| SRM | Study Reference Manual |
| SUSAR | Suspected unexpected serious adverse reactions |
| t1/2 | Apparent terminal phase half-life |
| tlag | Lag time for absorption |
| Tmax | Time of maximum observed concentration |
| TQT | Thorough QT |
| ULN | Upper limit of normal |
| VH | ViiV Healthcare |
| Vz/F | Apparent volume of distribution |
| WOCBP | Woman of childbearing potential |

## **Trademark Information**

| Trademarks of ViiV Healthcare |
|-------------------------------|
| NONE |

| Trademarks not owned by ViiV<br>Healthcare |
|--------------------------------------------|
| DAIDS |
| Phoenix WinNonlin |

## 10.2. Appendix 2: Clinical Laboratory Tests

- The tests detailed in Table 2 will be performed by the local laboratory.
- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Additional tests may be performed at any time during the study as determined necessary by the investigator or required by local regulations.
- Pregnancy Testing
  - Refer to Section 5.1 Inclusion Criteria for Screening pregnancy criteria.
  - Pregnancy testing (urine or serum as required by local regulations) should be conducted at the time points indicated in the SoA (Section 1.3).
  - Additional serum or urine pregnancy tests may be performed, as determined necessary by the investigator or required by local regulation, to establish the absence of pregnancy at any time during the participant's participation in the study.

 Table 2
 Protocol-Required Safety Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | |
|---|---|---|---|
| Hematology | Platelet Count Red Blood Cell Count | Red Blood Cell Indices: Mean corpuscular volume | White blood cell count with differential: Neutrophils |
| | Hemoglobin<br>Hematocrit | Mean corpuscular hemoglobin | Lymphocytes Monocytes Eosinophils Basophils Absolute neutrophil count |
| Clinical Chemistry 1 | Blood urea nitrogen Creatinine Glucose (fasting) Potassium Sodium Calcium Chloride Phosphorus | Carbon dioxide Aspartate aminotransferase Alanine aminotransferase Gamma-glutamyl transferase Total and direct bilirubin Lactate dehydrogenase Total cholesterol Triglycerides | Total protein Albumin Globulin Anion gap Alkaline phosphatase Uric acid Creatine phosphokinase Serum lipase Serum amylase |
| Routine Urinalysis | <ul> <li>Specific gravity</li> <li>pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase by dipstick</li> <li>Microscopic examination (if blood, leukocyte esterase, or protein is abnormal)</li> </ul> | | |

| Laboratory<br>Assessments | Parameters |
|---|---|
| Other Screening<br>Tests | Serology: HIV-1 and -2 antigen/antibody immunoassay, hepatitis B surface antigen, hepatitis C antibody |
| | <ul> <li>Alcohol, cotinine, and drug screen (to include at minimum amphetamines,<br/>barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines)</li> </ul> |
| | Pregnancy <sup>2</sup> |

- Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are given in Section 7.1 and Appendix 5. All events of ALT ≥3 ULN and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).
- 2 Serum testing will be performed on Screening and on Day -1. At all other timepoints, local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.

# 10.3. Appendix 3: Contraceptive Guidance and Collection of Pregnancy Information

#### 10.3.1. Definitions

#### **Woman of Childbearing Potential**

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of study intervention, additional evaluation should be considered.

#### Women in the following categories are not considered WOCBP

- 1. Premenarchal
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy
  - Documented bilateral tubal ligation

For individuals with permanent infertility due to an alternate medical cause other than the above, (e.g., Müllerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

- 3. Postmenopausal female
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
  - A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than 1 FSH measurement (>40 IU/L or mIU/mL) is required.
  - Females on HRT and whose menopausal status is in doubt will be required to
    use one of the non-estrogen hormonal highly effective contraception methods
    if they wish to continue their HRT during the study. Otherwise, they must
    discontinue HRT to allow confirmation of postmenopausal status before
    study enrollment.

## CONTRACEPTIVES<sup>a</sup> ALLOWED DURING AND AFTER THE STUDY INCLUDE THE FOLLOWING:

- Highly Effective Methods<sup>b</sup> That Have Low User Dependency: Failure rate of <1% per year when used consistently and correctly.
  - Non hormonal Intrauterine device
  - Bilateral tubal occlusion
  - Vasectomized partner

Note: Vasectomized partner is a highly effective contraceptive method provided that the partner is the sole sexual partner of the woman of childbearing potential and the absence of sperm has been confirmed. The documentation on male sterility can come from the site personnel's: review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner. If not, an additional highly effective method of contraception should be used. Spermatogenesis cycle is approximately 90 days.

- For the 28 days after study exit, women may resume oral hormonal contraceptives but double barrier methods (a combination of male condom with either cervical cap, diaphragm, or sponge with spermicide) must be used in addition.
- Highly Effective Methods<sup>b</sup> That Are User Dependent: Failure rate of <1% per year when used consistently and correctly.
  - Sexual abstinence

Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

Note: Periodic abstinence (calendar, sympto-thermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method (LAM) are not acceptable methods of contraception

- a. Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for those participating in clinical studies.
- b. Failure rate of <1% per year when used consistently and correctly. Typical use failure rates differ from those when used consistently and correctly.

#### 10.3.1. Collection of Pregnancy Information

#### Female participants who become pregnant

- Investigator will collect pregnancy information on any female participant, who becomes pregnant while participating in this study.
- Information will be recorded on the appropriate form and submitted to GSK within 24 hours of learning of a participant's pregnancy.

- Participant will be followed to determine the outcome of the pregnancy. The investigator will collect follow up information on participant and neonate, which will be forwarded to GSK. Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date.
- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-study pregnancy which is considered reasonably related to the study intervention by the investigator, will be reported to VH/GSK as described in Appendix 6. While the investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.

Any female participant who becomes pregnant while participating will discontinue study intervention or be withdrawn from the study.

## 10.4. Appendix 4: Regulatory, Ethical, and Study Oversight Considerations

## 10.4.1. Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines
  - Applicable International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines
  - Applicable laws and regulations
- The protocol, protocol amendments, ICF, CIB, and other relevant documents (e.g., advertisements) must be submitted to an IRB/IEC by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
  - Providing oversight of the conduct of the study at the site and adherence to requirements of 21 Code of Federal Regulations, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

#### 10.4.2. Financial Disclosure

Investigators and sub-investigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 10.4.3. Informed Consent Process

• The investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.

- Participants must be informed that their participation is voluntary. Participants
  or their legally authorized representative will be required to sign a statement of
  informed consent that meets the requirements of 21 Code of Federal Regulations
  Part 50, local regulations, ICH guidelines, Health Insurance Portability and
  Accountability Act (HIPAA) requirements, where applicable, and the IRB/IEC
  or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.
- Participants who are rescreened are required to sign a new ICF.

The ICF may contain a separate section that addresses the use of remaining mandatory samples for optional exploratory research in accordance with SOP-GSKF-410. The investigator or authorized designee will explain to each participant the objectives of the exploratory research. Participants will be told that they are free to refuse to participate and may withdraw their consent at any time and for any reason during the storage period. A separate signature will be required to document a participant's agreement to allow any remaining specimens to be used for exploratory research. Participants who decline to participate will not provide this separate signature.

#### 10.4.4. Data Protection

- Participants will be assigned a unique identifier by the sponsor. Any participant records or datasets that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

## 10.4.5. Publication Policy

• The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

- The sponsor will comply with the requirements for publication of study results.
   In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

## 10.4.6. Dissemination of Clinical Study Data

- Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a VH/GSK site or other mutually-agreeable location.
- VH/GSK will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study participants, as appropriate.
- The procedures and timing for public disclosure of the protocol and results summary and for development of a manuscript for publication for this study will be in accordance with VH/GSK Policy.
- VH/GSK intends to make anonymized patient-level data from this study available to external researchers for scientific analyses or to conduct further research that can help advance medical science or improve patient care. This helps ensure the data provided by study participants are used to maximum effect in the creation of knowledge and understanding.

## 10.4.7. Data Quality Assurance

- All participant data relating to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- Monitoring details describing strategy (e.g., risk-based initiatives in operations and quality such as Risk Management and Mitigation), methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the Monitoring Plan.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.

• The sponsor assumes accountability for actions delegated to other individuals (e.g., contract research organizations).

**CONFIDENTIAL** 

- Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICF, pertaining to the conduct of this
  study must be retained by the investigator for 25 years from the issue of the final
  Clinical Study Report/equivalent summary unless local regulations or
  institutional policies require a longer retention period. No records may be
  destroyed during the retention period without the written approval of the
  sponsor. No records may be transferred to another location or party without
  written notification to the sponsor.

#### 10.4.8. Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data reported on the CRF or entered in the electronic CRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.
- Definition of what constitutes source data can be found in the SRM.

## 10.4.9. Study and Site Closure

VH/GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of VH/GSK. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study intervention development

# 10.5. Appendix 5: Liver Safety: Required Actions and Follow-up Assessments

| Liver Chemistry Stopping Criteria | | |
|---|---|---|
| ALT-absolute | ALT ≥3 × ULN If ALT≥3 × ULN <b>AND</b> bilirubin <sup>1,2</sup> ≥2 × ULN (>35% direct bilirubin) or international normalized ratio (INR) >1.5, Report as an SAE. See additional Actions and Follow-Up Assessments listed below | |
| Required Actions and Follow up Assessments | | |
| Actions | | Follow-Up Assessments |
| <ul> <li>Report the event of the expectation o</li></ul> | AND bilirubin ≥2 × ULN or chemistries (include ALT, isaminase [AST], alkaline bilirubin and INR) and perform ow-up assessments within ipant twice weekly until liver esolve, stabilize or return to ee r hepatology consultation is | <ul> <li>Viral hepatitis serology³</li> <li>Obtain INR and recheck with each liver chemistry assessment until the transaminase values show downward trend</li> <li>Obtain blood sample for PK analysis, obtained within 48 hours of last dose⁴</li> <li>Serum CPK and lactate dehydrogenase.</li> <li>Fractionate bilirubin, if total bilirubin ≥2 × ULN</li> <li>Obtain complete blood count with differential to assess eosinophilia</li> <li>Record the appearance or worsening of clinical symptoms of liver injury, or hypersensitivity, on the AE report form</li> <li>Record use of concomitant medications on the concomitant medications report form including acetaminophen, herbal remedies, other over the counter medications.</li> <li>Record alcohol use on the liver event alcohol intake case report form</li> </ul> |
| If ALT ≥3 × ULN AND bilirubin <2 × ULN and INR ≤1.5: | | If ALT ≥3 × ULN AND bilirubin ≥2 × ULN or INR >1.5: |
| · | hemistries (include ALT, AST, ohatase, bilirubin and INR) and | Anti-nuclear antibody, anti-smooth muscle antibody, Type 1 anti-liver kidney |

## **Liver Chemistry Stopping Criteria**

perform liver event follow-up assessments within **24-72 hours** 

 Monitor participant weekly until liver chemistries resolve, stabilize or return to within Baseline

- microsomal antibodies, and quantitative total immunoglobulin G or gamma globulins.
- Serum acetaminophen adduct high performance liquid chromatography assay (quantifies potential acetaminophen contribution to liver injury in participants with definite or likely acetaminophen use in the preceding week [James, 2009]. NOTE: not required in China.
- Liver imaging (ultrasound, magnetic resonance, or computerized tomography) and /or liver biopsy to evaluate liver disease; complete Liver Imaging and/or Liver Biopsy CRF forms.
- Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation is not immediately available, discontinue study intervention for that participant if ALT ≥3 × ULN and bilirubin ≥ 2 × ULN. Additionally, if serum bilirubin fractionation testing is unavailable, record presence of detectable urinary bilirubin on dipstick, indicating direct bilirubin elevations and suggesting liver injury.
- 2. All events of ALT ≥3 × ULN and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and INR >1.5, which may indicate severe liver injury (possible "Hy's Law"), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis); the INR threshold value stated will not apply to participants receiving anticoagulants.
- 3. Includes: hepatitis A immunoglobulin (IgM) antibody, hepatitis B surface antigen, and hepatitis B core antibody; hepatitis C RNA; cytomegalovirus IgM antibody; Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, obtain heterophile antibody or monospot testing) and hepatitis E IgM antibody
- 4. Pharmacokinetic sample may not be required for participants known to be receiving placebo or non-GSK comparator interventions. Record the date/time of the PK blood sample draw and the date/time of the last dose of study intervention prior to PK blood sample draw on the CRF. If the date or time of the last dose is unclear, provide the participant's best approximation. If the date/time of the last dose cannot be approximated OR a PK sample cannot be collected in the time period indicated above, do not obtain a PK sample. Instructions for sample handling and shipping are in the SRM.

# 10.6. Appendix 6: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.6.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., ECG, radiological scans, vital signs measurements), including those that worsen from Baseline, considered clinically significant in the medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that

leads to the procedure is the AE.

- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.6.2. Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

#### A SAE is defined as any untoward medical occurrence that, at any dose:

#### Results in death

#### Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

## Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a pre-existing condition that did not worsen from Baseline is not considered an AE.

#### Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### Is a congenital anomaly/birth defect

#### Other situations:

• Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent 1 of the other outcomes listed in the above definition. These events should usually be considered serious.

Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## 10.6.3. Recording and Follow-Up of AE and SAE

#### AE and SAE Recording

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE/SAE information in the CRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to VH/GSK in lieu of completion of the GSK AE/SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by VH/GSK. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to VH/GSK.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### Assessment of Intensity

The investigator will make an assessment of intensity for each AE and SAE reported during the study using the DAIDS grading table Version 2.1, July 2017 (https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf) and assign it to 1 of the following categories:

- Mild: no or minimal interference with usual social and functional activities
- Moderate: greater than minimal interference with usual social and functional activities
- Severe: inability to perform usual social and functional activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized

for rating the intensity of an event; and both AE and SAE can be assessed as severe.

• Life Threatening: inability to perform basic self-care functions

An event is defined as "serious" when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the CIB and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to VH/GSK. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to VH/GSK.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is 1 of the criteria used when determining regulatory reporting requirements.

## Follow-up of AE and SAE

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by VH/GSK to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide VH/GSK with a copy of any

- postmortem findings including histopathology.
- New or updated information will be recorded in the originally completed CRF.
- The investigator will submit any updated SAE data to VH/GSK within 24 hours of receipt of the information.

## 10.6.4. Reporting of SAE to VH/GSK

#### SAE Reporting to VH/GSK via Electronic Data Collection Tool

- The primary mechanism for reporting SAE to VH/GSK will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) in order to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as it becomes available.
- The investigator or medically-qualified sub-investigator must show evidence within the electronic CRF (e.g., check review box, signature, etc.) of review and verification of the relationship of each SAE to study intervention/study participation (causality) within 72 hours of SAE entry into the electronic CRF.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section) or to the medical monitor by telephone.
- Contacts for SAE reporting can be found in the SRM.

## SAE Reporting to VH/GSK via Paper CRF

- Facsimile transmission of the SAE paper CRF is the preferred method to transmit this information to the medical monitor.
- In rare circumstances and in the absence of facsimile equipment, notification by telephone is acceptable with a copy of the SAE data collection tool sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE CRF pages within the designated reporting time frames.
- Contacts for SAE reporting can be found in SRM.

## 10.7. Appendix 7: Genetics

#### **USE/ANALYSIS OF DNA**

- Genetic variation may impact a participant's response to study intervention, susceptibility, severity, and progression of disease. Variable response to study intervention may be due to genetic determinants that impact drug absorption, distribution, metabolism, and excretion; mechanism of action of the drug; disease etiology; and/or molecular subtype of the disease being treated. Therefore, where local regulations and IRB/IEC allow, a blood sample will be collected for DNA analysis.
- DNA samples will be used for research related to GSK3640254 or HIV and related diseases. They may also be used to develop tests/assays including diagnostic tests related to GSK3640254 or HIV MIs and HIV. Genetic research may consist of the analysis of 1 or more candidate genes or the analysis of genetic markers throughout the genome or analysis of the entire genome (as appropriate).
- DNA samples will be analyzed if it is hypothesized that this may help further understand the clinical data.
- The samples may be analyzed as part of a multi-study assessment of genetic factors involved in the response to GSK3640254 or study interventions of this class. The results of genetic analyses may be reported in the clinical study report or in a separate study summary.
- The sponsor will store the DNA samples in a secure storage space with adequate measures to protect confidentiality.
- The samples will be retained while research on GSK3640254 (or study interventions of this class) or HIV continues but no longer than 15 years after the last participant's last visit or other period as per local requirements.

#### 11. REFERENCES

Bristol-Myers Squibb Company Document Control Number 930109388. A randomized, double-blind, double-dummy, positive-controlled, crossover study to determine electrocardiographic effects of BMS-955176 in healthy subjects. Report Date: 13 January 2017.

Department of Health and Human Services (DHHS), Food and Drug Administration, Center for Drug Evaluation and Research (US). Guidance for Industry: Food-Effect Bioavailability and Fed Bioequivalence Studies. December 2002 [12 screens]. Available from:

http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM070241.pdf

GlaxoSmithKline Document Number 2016N302783\_00. Clinical Study Report: A Phase 2b Randomized, Active-Controlled, Double-Blind Trial to Investigate Safety, Efficacy and Dose-response of BMS-955176/GSK3532795, Given on a Backbone of Tenofovir/Emtricitabine, in Treatment-Naive HIV-1 Infected Adults – Week 24 Interim Analysis, 21 Jun 2017.

GlaxoSmithKline Document Number 2017N322200\_00. A Phase 2b Randomized, Active-Controlled, Staged, Open-Label Trial to Investigate Safety and Efficacy of BMS-955176/GSK3532795 in Combination with Dolutegravir and Atazanavir (with or without Ritonavir) in Treatment-Experienced HIV-1 Infected Adults. 25 September 2018.

GlaxoSmithKline Document Number 2018N375461\_00. Clinical Pharmacology Synopsis. A Double-Blind (Sponsor Unblinded), Randomized, Placebo-Controlled, Single and Repeated Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK3640254 in Healthy Participants. September 2018.

GlaxoSmithKline Document Number 2018N379610\_00. GSK3640254 Investigator's Brochure, Version 01. Effective Date: 04 Oct 2018.

Hasler WL. Nausea, Vomiting, and Indigestion: Introduction. Chapter 39. Harrisons Principles of Internal Medicine 18th edition. 2012. McGraw Hill.

James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, et al. Pharmacokinetics of acetaminophen - protein adducts in adults with acetaminophen overdose and acute liver failure. Drug Metab Disp. 2009;37(8):1779-84.

Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007;164(7):1035-43.

Rome Foundation. Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders. Available:

http://www.theromefoundation.org/assets/pdf/19\_RomeIII\_apA\_885-898.pdf. Accessed 18 Feb 2019.

Soll AH and Graham DY. Peptic Ulcer Disease. Chapter 40. Textbook of Gastroenterology. 5th edition. 2009. Blackwell Publishing.